CLINICAL TRIAL: NCT00018967
Title: A Trial of Carboxypeptidase-G2 (CPDG2) For The Management of Patients With Intrathecal Methotrexate Overdose
Brief Title: Carboxypeptidase-G2 in Treating Nervous System Toxic Effects in Patients Given an Overdose of Intrathecal Methotrexate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Oncology Group (Network)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000077521; NCI-92-C-0137N; CCG-0923; POG-9688; NCI-T92-0021N; COG-0923; COG-P9688; NCT00001299 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Neurotoxicity; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific; neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — glucarpidase

INTERVENTIONS:
Drug: glucarpidase

SUMMARY:
RATIONALE: Chemoprotective drugs such as carboxypeptidase-G2 may protect normal cells from the toxic effects of chemotherapy.

PURPOSE: Clinical trial to study the effectiveness of carboxypeptidase-G2 in treating nervous system toxic effects in patients given an accidental overdose of intrathecal methotrexate.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of carboxypeptidase-G2 rescue in patients who develop life threatening methotrexate (MTX) neurotoxicity following accidental intrathecal MTX overdose.
* Study the CSF pharmacokinetics of MTX following rescue.

OUTLINE: Patients undergo a lumbar puncture as soon as possible after methotrexate overdose to remove methotrexate and receive a single dose of carboxypeptidase-G2 intrathecally over 5 minutes.

Patients are followed for at least 1 month.

PROJECTED ACCRUAL: A maximum of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients who received an intrathecal overdose of methotrexate of 100 mg or more

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior anaphylactic reaction to carboxypeptidase-G2 administration

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Concurrent therapy allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 1993-11; Primary Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C. Widemann, MD, Study Chair — National Cancer Institute (NCI)
Locations (103):
- United States (88):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center at UV Health System, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- Swiss Pediatric Oncology Group Geneva, Geneva, Switzerland

REFERENCES:
- [Result] Widemann BC, Balis FM, Shalabi A, Boron M, O'Brien M, Cole DE, Jayaprakash N, Ivy P, Castle V, Muraszko K, Moertel CL, Trueworthy R, Hermann RC, Moussa A, Hinton S, Reaman G, Poplack D, Adamson PC. Treatment of accidental intrathecal methotrexate overdose with intrathecal carboxypeptidase G2. J Natl Cancer Inst. 2004 Oct 20;96(20):1557-9. doi: 10.1093/jnci/djh270. PMID 15494606
- [Result] Widemann BC, Balis FM, Shalabi A, et al.: Carboxypeptidase-G2 (CPDG2) treatment of accidental intrathecal (IT) methotrexate (MTX) overdose. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-490, 2002.